CLINICAL TRIAL: NCT01033773
Title: STEP-DC: Stop Emergency Room Visits for Uncontrolled Hyperglycemia Project in the District of Columbia
Brief Title: Stop Emergency Room Visits for Hyperglycemia Project - District of Columbia (DC)
Acronym: STEP-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Michelle Magee, Director, MedStar Diabetes Institute, Medstar Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-268
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Uncontrolled hyperglycemia; Emergency Department
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes education and medication management (Other): All enrolled patients received the intervention. There was no comparative arm. The analysis was done as pre and post.
  Interventions: Drug: Antihyperglycemic medication guideline for management of uncontrolled hyperglycemia presenting to the ED using metformin, sulfonylurea and/or insulin; Behavioral: Diabetes survival skills self-management education

INTERVENTIONS:
Drug: Antihyperglycemic medication guideline for management of uncontrolled hyperglycemia presenting to the ED using metformin, sulfonylurea and/or insulin — Diabetes medications (including sulfonylureas, metformin and/or insulin) were initiated and/or adjusted at each visit using the intervention algorithm per presenting blood glucose and prior diabetes medications.
Behavioral: Diabetes survival skills self-management education — Survival skills DSME based upon current JCAHO and ADA joint recommendations for persons with diabetes prior to discharge to the outpatient setting was initiated in the ED and continued at the follow-up encounters.

SUMMARY:
To demonstrate that a focused Emergency Department (ED) intervention for uncontrolled hyperglycemia enables safe and effective glycemic management and reduces emergency room re-visits. We assessed hypoglycemia BG < 60mg/dL; change in mean blood glucose and A1C, and ED revisits for hyperglycemia.

DETAILED DESCRIPTION:
Patients with BG > 200mg/dL presenting to an urban tertiary care hospital ED were enrolled in a 4 week prospective intervention with historic self-controls. Subjects returned at 12-72 hours, 2 and 4 weeks. Diabetes medications (including sulfonylureas, metformin and/or insulin) were initiated and/or adjusted at each visit using the intervention algorithm per presenting blood glucose and prior diabetes medications. Survival skills self-management education and navigation to outpatient services were provided.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type 2 Diabetes Mellitus,
* random BG > 200 mg/dL,
* willing and able to provide informed consent and to participate in diabetes self-management education (DSME)
* stable for discharge from the ED once hyperglycemia treatment initiated.

Exclusion Criteria:

* type 1 Diabetes Mellitus,
* diabetic ketoacidosis or hyperosmolar non-ketotic state,
* concomitant treatment with glucocorticoids (other than stable maintenance dose therapy),
* cognitive or physical impairment preventing participation in DSME
* unwillingness or inability to provide consent and/or attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Magee, MD, MBBCh, Principal Investigator — Medstar Diabetes and Research Institutes, Georgetown University School of Medicine.
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Education and Medication Management
Started | 86
Completed | 51
Not Completed | 35

BASELINE CHARACTERISTICS:
Groups:
- Intervention: All enrolled patients received the intervention. There was no comparative arm. The analysis was done as pre and post.
  Antihyperglycemic medication guideline for management of uncontrolled hyperglycemia presenting to the ED using metformin, sulfonylurea and/or insulin: Diabetes medications (including sulfonylureas, metformin and/or insulin) were initiated and/or adjusted at each visit using the intervention algorithm per presenting blood glucose and prior diabetes medications.
  Diabetes survival skills self-management education: Survival skills DSME based upon current JCAHO and ADA joint recommendations for persons with diabetes prior to discharge to the outpatient setting was initiated in the ED and continued at the follow-up encounters.
Arm/Group | Intervention
Number analyzed (Participants) | 86
Age, Customized [Count of Participants; unit: Participants]
  Age 18-44 | 28
  Age 45-64 | 51
  Age 65 and older | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 76
  White | 4
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Hypoglycemia Events (Blood Glucose < 60mg/dL) Within 24 Hours of Baseline Visit
Description: Total Number of hypoglycemic events defined as Blood Glucose < 60 within 24 hours of index emergency room visit (baseline)
Time Frame: 24 hours
Measure: Number; unit: events
Arm/Group | Intervention
Number analyzed (Participants) | 86
events | 0

2. Secondary Outcome: Change in Mean Blood Glucose From Time of Presentation to Emergency Room to End of Intervention 30 Days From Baseline
Description: Mean difference in of blood glucose in mg/dl between baseline mean BG and end of intervention mean BG 30 days from baseline
Time Frame: 30 days
Population: This data was only available for 51 patients therefore only 51 patients' results were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intervention
Number analyzed (Participants) | 51
mg/dl
  Mean BG at baseline | 356 (110)
  Mean BG at end of intervention | 183 (103)

3. Secondary Outcome: Change in Hemoglobin A1C From Baseline to End of Intervention at 30 Days
Description: difference between mean hemoglobin A1C at baseline and mean Hemoglobin A1C to end of intervention
Time Frame: 30 days
Population: Only 46 patients had a baseline and end of intervention A1C available therefore only 46 participants are included in the data
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin A1C
Arm/Group | Intervention
Number analyzed (Participants) | 46
percentage of hemoglobin A1C
  Mean baseline A1C | 12.0 (1.5)
  Mean end of intervention A1C | 11.6 (1.6)

ADVERSE EVENTS:
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 14/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=86)
Hypoglycemia (Endocrine disorders) | 14 (26) — Blood sugar less then 70 mg/dl

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes